CLINICAL TRIAL: NCT02664818
Title: China Heart Failure Registry Study: A Multicenter, Prospective Investigation of Clinical Characteristics, Treatment, and Outcome of Patients Hospitalized With Heart Failure
Brief Title: Study of China Heart Failure Registry to Investigate Characteristics of Patients in China
Acronym: China-HF
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chinese Academy of Medical Sciences, Fuwai Hospital (Other)
Responsible Party: Principal Investigator, Jian Zhang, Director of Heart Failure Center, Fuwai hospital; vice-chairmen of Chinese Heart Failure Association, Chinese Academy of Medical Sciences, Fuwai Hospital
Other Study IDs: 2011BA111B02
Record Dates: First submitted 2016-01-11; First posted 2016-01-27 (Estimated); Last update posted 2016-01-27 (Estimated); Status verified 2016-01

CONDITIONS: Heart Failure
Keywords: Heart failure; China; Registry; Characteristic; Outcome
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Heart failure: Hospitalized patients with primary discharge diagnosis of heart failure and who were aged 18 years or older.

SUMMARY:
The purpose of this study is to assess clinical characteristics, treatment, and outcome of patients hospitalized with heart failure in China and compared those with other registries

DETAILED DESCRIPTION:
* All sites were monitored randomly every year. Trained monitors were designated to monitor the process, compliance of enrollment criteria and accuracy of original data by visiting every site.
* In order to make sure the accuracy of data collected, we make some restrictions (range or format) and reminding functions in the electronic Case Report Form (eCRF).
* Detail information of each variable has been pre-defined. Staffs were trained before data entry.
* Standard Operating Procedures: Case data were collected by printed Case Report Form (CRF) and entered into a web-based data center (http://103.31.202.60/subFW/). Hospitals that did not complete eCRF would send printed CRF to data center. Trained clinicians or staffs were asked to enter these data into the web-based eCRF. Following variables were included in the database: (i) demography and characteristics of patients: age, gender, medical history, life style, precipitating factors of HF, laboratory tests, ECG, chest X-ray and comorbidities diagnosed at discharge. Physical examination, echocardiography, laboratory tests were performed at both admission and discharge; (ii) Heart failure management included pharmacological treatments (before admission, during hospitalization and at discharge), and nonpharmacological treatments (including coronary revascularization, implantable cardioverter-defibrillator, cardiac resynchronization therapy, pacemakers, and surgical or transcatheter valvular therapies, electrical conversion, intra aortic balloon pump, continuous renal replacement therapy, and invasive mechanical ventilation).The causes of in-hospital death included sudden death, cardiac death and non-cardiac death. All patients were followed up after discharge in outpatient department, or via electronic hospital records, or conversations with patients or patients' families by telephone. Outcomes for post-discharge included death (sudden death, cardiac death and non-cardiac death), and rehospitalization for heart failure deterioration, acute coronary syndrome, cardiac shock, syncope, and cardiac transplantation were recorded and entered into the web-based database. Information about physical examination, laboratory tests, ECG, chest X-ray, echocardiography, and costs and use of medications were collected at each follow-up visit.
* Sample size: A total of 15000 patients with heart failure were planned to be recruited from hospitals based on classification of economic-geographic regions in China, and a minimum number of patients were expected to enroll according to the number of hospitalized cases for each hospital. By September 2015, data from 13687 patients have been collected.
* Plan for missing data: Validated data was used to describe the clinical characteristics and treatment of patients without considering those missing. As for September 2015, the missing data on most of variables accounts for no more than 10% of all patients (n = 13687). Furthermore, variables obtained in multiple Logistic regression models (10318) for death were from over three quarters of (75.4%) of all patients. Simple and multiple imputation methods were not used in this study because of a large number of patients has been validated for analysis.
* Statistical analysis plan: Clinical characteristics, treatments, and outcomes were described by using means ± standard deviation or interquartile range (IQR) for continuous variables, and absolute numbers and percentages for categorical variables. The comparison of subgroups were performed by Student t-test or ANOVA for symmetrical continuous, Mann-Whitney U or Kruskal-Wallis H test for nonsymmetric continuous, and χ2 tests for categorical variables. Logistic regression was used to select potential risk factors for outcomes. Candidate variables associated with mortality in univariable Logistic regression analysis (P ≤ 0.20) were proceeded with multivariable analysis. Variables with significant P values (P < 0.05) were retained in the final multivariable model. Logarithmic transformation was performed to normalize the distribution of variables with skewed distribution. All P values of less than 0.05 from two-sided tests were accepted as statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized patients with primary discharge diagnosis of heart failure according to current Chinese Heart Failure Guideline were recruited from January 2012.

Exclusion Criteria:

* Hospitals were excluded if they declined to participate or did not admit patients with heart failure.No other exclusion criteria were defined.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients hospitalized with primary discharge diagnosis of heart failure
Sampling Method: Non-Probability Sample
Enrollment: 15000 (Estimated)
Dates: Start 2012-01; Primary Completion 2016-04 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
The overall composite of 9 performance measures for heart failure medications compliance. | Duration of hospital stay, an expected average of 10 days
  1. Prescribed rate of ACEIs/ARBs in patients with acute decompensated heart failure (ADHF) before admission.
  2. Prescribed rate of β blockers in patients with ADHF before admission.
  3. Prescribed rate of diuretics in patients with ADHF before admission.
  4. Prescribed rate of aldosterones in patients with ADHF before admission.
  5. Prescribed rate of ACEIs/ARBs in appropriate patients discharged alive.
  6. Prescribed rate of β blockers in appropriate patients discharged alive.
  7. Prescribed rate of diuretics in all patients discharged alive.
  8. Prescribed rate of aldosterones in appropriate patients discharged alive.
  9. Prescribed rate of warfarins in patients with nonvalvular atrial fibrillation and CHA2DS2-VASc score ≥2 discharged alive.

SECONDARY OUTCOMES:
Number of deaths during index of hospitalization and after discharge. | Duration of hospital stay with an expected average of 10 days for in-hospital death; 1 year for patients discharged alive

CONTACTS AND LOCATIONS:
Overall Officials: Jian Zhang, Ph. D, Study Chair — Fuwai Hospital, National Center for Cardiovascular Diseases, Chinese Academy of Medical Sciences and Peking Union Medical College
Locations (1):
- Fuwai Hospital, National Center for Cardiovascular Diseases, Chinese Academy of Medical Sciences and Peking Union Medical College, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
Data were abstracted by printed Case Report Form and entered into a web-based data center (http://103.31.202.60/subFW/). Hospitals that did not complete electronic CRF (eCRF) would send printed CRF to data center. Trained clinicians or staffs would enter these data into web-based eCRF.

REFERENCES:
- [Derived] Wu Y, Zhang Y, Zhang J. Low Aortic Pulsatility Index and Pulmonary Artery Pulsatility Index Are Associated With Increased Mortality in Patients With Dilated Cardiomyopathy Awaiting Heart Transplantation. Korean Circ J. 2025 Feb;55(2):134-147. doi: 10.4070/kcj.2024.0192. Epub 2024 Oct 17. PMID 39506184
- [Derived] Huang BP, Zhao L, Zhao XM, Zhai M, Huang Y, Zhou Q, Tian PC, Liang L, Huang LY, Feng JY, Zhang YH, Zhang J. Serum Potassium Levels and Mortality in Hospitalized Heart Failure Patients. Rev Cardiovasc Med. 2023 Aug 9;24(8):228. doi: 10.31083/j.rcm2408228. eCollection 2023 Aug. PMID 39076700
- [Derived] Huang B, Huang Y, Zhai M, Zhou Q, Ji S, Liu H, Zhuang X, Zhang Y, Zhang J. Association of Sex With Cardiovascular Outcomes in Heart Failure Patients With Obstructive or Central Sleep Apnea. J Am Heart Assoc. 2024 Mar 5;13(5):e031186. doi: 10.1161/JAHA.123.031186. Epub 2024 Feb 27. PMID 38410942
- [Derived] Wu Y, Tian P, Liang L, Chen Y, Feng J, Huang B, Huang L, Zhao X, Wang J, Guan J, Li X, Zhang Y, Zhang J. Afterload-related cardiac performance is a powerful hemodynamic predictor of mortality in patients with chronic heart failure. Ther Adv Chronic Dis. 2023 Jun 5;14:20406223231171554. doi: 10.1177/20406223231171554. eCollection 2023. PMID 37324410
- [Derived] Zhao L, Zhao X, Tian P, Liang L, Huang B, Huang L, Feng J, Zhang Y, Zhang J. Predictive value of remnant cholesterol level for all-cause mortality in heart failure patients. Front Cardiovasc Med. 2023 Feb 15;10:1063562. doi: 10.3389/fcvm.2023.1063562. eCollection 2023. PMID 36873397
- [Derived] Liang L, Zhao X, Huang L, Tian P, Huang B, Feng J, Zhou P, Wang J, Zhang J, Zhang Y. Prevalence and prognostic importance of malnutrition, as assessed by four different scoring systems, in elder patients with heart failure. Nutr Metab Cardiovasc Dis. 2023 May;33(5):978-986. doi: 10.1016/j.numecd.2023.01.004. Epub 2023 Jan 11. PMID 36710105
- [Derived] Zhao L, Zhao X, Tian P, Liang L, Huang B, Huang L, Feng J, Zhang Y, Zhang J. Prognostic utility of the prognostic nutritional index combined with serum sodium level in patients with heart failure. Nutr Metab Cardiovasc Dis. 2022 Aug;32(8):1894-1902. doi: 10.1016/j.numecd.2022.04.004. Epub 2022 Apr 14. PMID 35637081
- See also: Data were abstracted by electronic form created in this web site — http://103.31.202.60/subFW/